CLINICAL TRIAL: NCT02469272
Title: Fecal Microbiota Transplantation (FMT) in Nonalcoholic Steatohepatitis(NASH). A Pilot Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Kittichai Promrat, M.D., Associate Professor, Lifespan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Committee # 2014-15
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Intervention: standardized preparation of frozen fecal material from lean healthy donors Route: infused into the duodenum through the working channel of the instrument at upper endoscopy Dosing: 1 dose
  Interventions: Drug: Fecal Microbiota Transplantation

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Administration of frozen fecal materials into gastrointestinal tract
  Other Names: FMT

SUMMARY:
Nonalcoholic steatohepatitis (NASH) is common, may progress to cirrhosis and is predicted to become a leading indication for liver transplantation in the near future. Though often associated with obesity and the metabolic syndrome, our current understanding of disease development is limited and there are few therapeutic options. Imbalance of gut bacteria is suspected to play a key role driving the progression of fatty liver disease and there is hope manipulation of these bacteria may be beneficial. This study will determine if fecal microbiota transplantation, using stool from lean donors, is an effective and safe treatment for NASH.

DETAILED DESCRIPTION:
Nonalcoholic Steatohepatitis (NASH), a severe form of fatty liver disease, is highly prevalent and can lead to cirrhosis, liver failure and hepatocellular carcinoma. It is strongly associated with obesity and the metabolic syndrome. The impact of the gut microbiota on obesity and the metabolic syndrome is potentially large and increasing evidence suggests that dysbiosis might contribute to the development of NASH. There is a fundamental gap in understanding how alterations in the intestinal microbiota lead to a wide range of metabolic syndrome associated conditions including fatty liver disease in humans. The long-term goal of this project is to better understand the mechanisms linking intestinal dysbiosis and extra-intestinal clinical phenotypes, in particular obesity and NAFLD. Compositional shifts in gut bacteria from antibiotic use can perpetuate diseases such as Clostridum difficile infection, and manipulation of the microbiota through stool transplant from healthy donors can be used to cure disease. The objective of this application is to determine whether restoration of beneficial gut microbiota via fecal microbiota transplantation using stool from lean donors (FMT-L) improves NASH. The central hypothesis for this project is that transfer of gut microbiota from lean donors will result in reduced hepatic steatosis, and improved histological and biochemical features of NASH, all of which will correlate with observed changes in the small bowel and distal gut microbiome. This hypothesis will be tested by pursuing 3 specific aims: 1) determine the effect of FMT-L in patients with NASH on hepatic steatosis and markers of NASH; 2) perform microbiome analyses on pre- and post-FMT-L small bowel & stool samples; and 3) investigate mechanistic correlates linking dysbiosis with histologic changes in NASH after FMT-L. The study will be a pilot open labeled trial examining the effect of FMT-L in patients with biopsy proven NASH. The primary outcome measure will be a change in MRI-determined hepatic fat fraction,12 weeks after transplantation. Differences in the microbiota after FMT-L in the small bowel and distal gut, including the durability of microbiota changes, will be examined using advanced metagenomic techniques. Clinical and laboratory features of the metabolic syndrome and obesity as well as hepatic and systemic inflammatory markers will be examined for mechanistic correlates linking dysbiosis with histologic changes in the liver. In addition to understanding how the gut microbiota affects fatty liver disease progression, study findings will provide a framework for future microbiome research on metabolic syndrome related diseases such as diabetes, obesity, and other inflammatory disorders. An increased understanding of how the human gut microbiota is altered in metabolic disease may open a new avenue of therapeutics based on manipulation of gut bacteria.

ELIGIBILITY:
Inclusion Criteria:

1) >18 years of age 2) histologic evidence of definite or probable NASH based upon a liver biopsy obtained <90 days prior to enrollment and a NAFLD activity score (NAS) ≥4 with ≥1 in each component of the NAS score (steatosis, scored 0-3, ballooning degeneration, 0-2, and lobular inflammation, 0-3).

-

Exclusion Criteria:

1. current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 g/day in females and more than 30 g/day in males, on average)
2. Another form of liver disease
3. Recent antibiotic use within 3 months or need for chronic antibiotic therapy
4. Use of drugs historically associated with NAFLD or drugs known to improve NASH histology such as vitamin E> 400 IU/day or pioglitazone
5. Prior or planned (during the study period) bariatric surgery
6. Uncontrolled diabetes defined as HbA1c 9.5% or higher within 60 days prior to enrollment
7. Presence of cirrhosis on liver biopsy
8. Clinical evidence of hepatic decompensation
9. Inability to safely obtain a liver biopsy or perform an upper endoscopy
10. Human Immunodeficiency Virus (HIV) infection
11. Active, serious medical disease with likely life expectancy less than 5 years
12. Active substance abuse including inhaled or injection drugs in the year prior to screening
13. pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial, breast feeding
14. Participation in an IND trial in the 30 days before randomization
15. Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study
16. History of severe (anaphylactic) food allergy
17. History of inflammatory bowel disease
18. History of gastroparesis or altered gastric motility -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
degree of hepatic steatosis as determined by MRI | 12 weeks

SECONDARY OUTCOMES:
Liver Function Tests | 12 weeks
Markers of insulin sensitivity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kittichai Promrat, M.D., Principal Investigator — Lifespan; Colleen Kelly, M.D., Principal Investigator — Lifespan
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Kelly CR, Ihunnah C, Fischer M, Khoruts A, Surawicz C, Afzali A, Aroniadis O, Barto A, Borody T, Giovanelli A, Gordon S, Gluck M, Hohmann EL, Kao D, Kao JY, McQuillen DP, Mellow M, Rank KM, Rao K, Ray A, Schwartz MA, Singh N, Stollman N, Suskind DL, Vindigni SM, Youngster I, Brandt L. Fecal microbiota transplant for treatment of Clostridium difficile infection in immunocompromised patients. Am J Gastroenterol. 2014 Jul;109(7):1065-71. doi: 10.1038/ajg.2014.133. Epub 2014 Jun 3. PMID 24890442
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514